CLINICAL TRIAL: NCT06771219
Title: A Phase 1 Dose-Escalation Study of SLV-154 in Subjects With Metastatic Solid Tumors
Brief Title: SLV-154 Treatment of Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Solve Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLV-154-01Tx
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Cancer of Head and Neck (SCCHN); NSCLC; SCLC; Cervical Cancer Metastatic; Breast Cancer Metastatic; Endometrial Cancer; Ovarian Cancer; Urothelial Cancer; Sarcoma; Thyroid Cancer
Keywords: metastatic solid tumors; metastatic cancer; solid tumor
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Sarcoma; Thyroid Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: In this study, a BOIN design with a target DLT rate for the MTD of 27% and an estimated maximum sample size of ~70 subjects will be used to guide the dose escalation and determine the RDR of SLV-154.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Level 1 (Experimental): 0.75 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 2 (Experimental): 1.5 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 3 (Experimental): 3.0 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 4 (Experimental): 5.0 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 5 (Experimental): 7.5 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 6 (Experimental): 10.0 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 7 (Experimental): 12.5 mg/kg
  Interventions: Drug: SLV-154
- Dose Level 8 (Experimental): 15.0 mg/kg
  Interventions: Drug: SLV-154

INTERVENTIONS:
Drug: SLV-154 — SLV-154

SUMMARY:
This is a Phase 1 dose-escalation study evaluating the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and efficacy of SLV-154 across a range of dose levels when administered to subjects with metastatic solid tumors.

DETAILED DESCRIPTION:
A Bayesian optimal interval (BOIN) design with a target dose-limiting toxicity (DLT) rate for the maximum tolerated dose (MTD) of 27% and an estimated maximum sample size of ~70 subjects will be used to guide the dose escalation and determine the recommended dosing regimen (RDR) of SLV-154.

SLV-154 will be administered intravenously (IV) in repeated 3-week cycles. Treatment will continue until progressive disease or discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women (as appropriate for cancer type) of age ≥18 years.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
3. Histologically or cytologically confirmed diagnosis of solid tumor as documented in medical records with the primary history comprising one of the following:

   1. SCCHN
   2. NSCLC
   3. SCLC
   4. Breast cancer
   5. Cervical cancer
   6. Endometrial cancer
   7. Ovarian cancer
   8. Urothelial cancer
   9. Sarcoma
   10. Thyroid cancer
4. Presence of metastatic disease that has progressed during or following previous treatment.
5. Presence of radiographically measurable disease.
6. Prior receipt of commercially available therapies that are indicated for the subject's cancer and have demonstrated survival benefit for that indication.
7. Availability of tumor tissue from a fresh tumor biopsy obtained by a core needle, excisional, or incisional biopsy; or punch biopsy (for cutaneous disease); or archival tumor sample from a previous biopsy.
8. Availability of computed tomography (CT) or magnetic resonance imaging (MRI) of chest, abdomen, and pelvis, and/or fluorodeoxyglucose (FDG) positron emission tomography (PET)/CT (if appropriate for tumor type) (with PET from base of the skull to mid-thigh, if performed) within 35 days before study drug administration.
9. Completion of all previous therapy (including surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy, or investigational therapy) for the treatment of cancer ≥1 week before the start of study drug administration.
10. Adequate hematological profile.
11. Adequate coagulation profile.
12. Adequate hepatic profile.
13. Adequate renal function.
14. Negative viral serology or adequate therapy for human immunodeficiency virus (HIV), hepatitis B (HBV), and hepatitis C (HCV) infection.
15. For female subjects of childbearing potential, a negative serum pregnancy test.
16. For female subjects of childbearing potential, willingness to use a protocol-recommended method of contraception from the start of the screening period until ≥6 months after the final dose of study therapy.
17. For male subjects who can father a child and are having intercourse with females of childbearing potential who are not using adequate contraception, willingness to use a protocol-recommended method of contraception from the start of study therapy until ≥6 months after the final dose of study therapy and to refrain from sperm donation from the start of study therapy until ≥12 months after administration of the final dose of study therapy.
18. Willingness and ability of the subject to comply with scheduled visits, the drug administration plan, protocol-specified laboratory tests, other study procedures (including required tumor biopsy/aspirations and/or radiographic studies), and study restrictions.
19. Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

1. Malignancy involving the central nervous system unless brain metastases have been previously treated with radiotherapy, have been stable for ≥4 weeks, and do not require corticosteroids.
2. Presence of another cancer with disease manifestations or therapy that could adversely affect subject safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results.
3. Uncontrolled ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infection) at the time of start of study therapy.
4. Significant cardiovascular event or comorbidity.
5. Significant screening ECG abnormalities.
6. Pregnancy or breastfeeding.
7. Major surgery within 4 weeks before the start of study therapy.
8. Use of a strong inhibitor or inducer of CYP3A4 or CYP1A2.
9. Use of a drug known to prolong the QT interval within 7 days prior to the start of study drug administration.
10. Concurrent participation in another therapeutic or imaging clinical trial.
11. Other conditions likely to interfere with a subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
MTD and/or RDR | Through the duration of treatment, up to approximately 18 months
  Determination of the MTD (maximum tolerated dose) and/or RDR (recommended dosing regimen) for SLV-154

SECONDARY OUTCOMES:
SLV-154 administration | Through the duration of treatment, up to approximately 18 months
  SLV-154 drug administration as assessed by prescribing records
SLV-154 Safety | Through the duration of treatment, up to approximately 18 months
  Collection of type, frequency, severity, timing of onset, duration, and relationship to study drug of any treatment-emergent adverse events (TEAEs); laboratory abnormalities; vital sign/oxygen saturation abnormalities; adverse electrocardiogram (ECG) findings; DLTs; serious adverse events (SAEs); adverse events of special interest (AESIs); or adverse events (AEs) leading to interruption, modification, or discontinuation of study drug administration.
Evaluation of use of concomitant medications | Through the duration of treatment, up to approximately 18 months
  Type, frequency, and timing of use of supportive care and other concomitant medications
SLV-154 Pharmacokinetics | Varying timepoints through the duration of treatment, up to approximately 18 months
  Evaluation of the pharmacokinetic profile of SLV-154
Immunogenicity | Varying timepoints through the duration of treatment, up to approximately 18 months
  Measurement of changes in titers of circulating SLV 154-reactive antibodies (as assessed using immunoassay methods)
Objective Response Rate (ORR) | Through the duration of treatment, up to approximately 18 months
  ORR assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria and defined as the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR).
Time to Response (TTR) | Up to approximately 36 months
  TTR: interval from the start of study drug administration to the first documentation of objective tumor regression
Duration of Response (DOR) | Up to approximately 36 months
  DOR: interval from the first documentation of objective tumor regression to the earlier of the first documentation of disease progression or death from any cause
Progression-free survival (PFS) | Up to approximately 36 months
  PFS: interval from the start of study drug administration to the earlier of the first documentation of disease progression or death from any cause
Time to treatment failure (TTF) | Up to approximately 36 months
  TTF: interval from the start of study drug administration to the earliest of the first documentation of disease progression, the permanent cessation of study drug due to an AE, or death from any cause
Overall survival (OS) | Up to approximately 36 months
  OS: interval from the start of study drug administration to death from any cause

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Washington University, St Louis, Missouri
  - Astera Cancer Care, East Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Mays Cancer Center; University of Texas Health San Antonio, San Antonio, Texas
  - University of Washington / Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
A CSR and publication of results is planned but we currently do not intend to share individual participant data with other researchers.